CLINICAL TRIAL: NCT04429243
Title: GORE® VIABAHN® Endoprosthesis Post-Marketing Surveillance Study - Treatment of Patients With Stenosis or Occlusion at the Venous Anastomosis of Synthetic Arteriovenous (AV) Access Graft
Brief Title: GORE® VIABAHN® Endoprosthesis Post-Marketing Surveillance Study
Status: Completed | Type: Observational
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Other Study IDs: JPS 19-05: AVR PMS
Record Dates: First submitted 2020-05-27; First posted 2020-06-12 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Vascular Stent-Graft Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GORE® VIABAHN® Stent Graft: Participants will be examined 1, 3, 6, 12 and 24 months following the GORE® VIABAHN® Stent Graft installation.
  Interventions: Device: GORE® VIABAHN® Stent Graft

INTERVENTIONS:
Device: GORE® VIABAHN® Stent Graft — On Day 1, participants will receive the GORE® VIABAHN® Stent Graft.

SUMMARY:
This study will confirm the efficacy and safety in the clinical setting after the launch of the GORE® VIABAHN® stent graft (hereafter referred to as "Viabahn") for the treatment of patients with stenosis or occlusion at the venous anastomosis of synthetic arteriovenous access graft.

ELIGIBILITY:
Inclusion Criteria:

* Participants who developed stenosis or occlusion at the venous anastomosis of synthetic arteriovenous access graft
* Participants who was used to repair vascular access circuits for purposes other than treatment of stenosis or occlusion at the venous anastomosis of synthetic arteriovenous access graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stenosis or occlusion at the venous anastomosis of synthetic arteriovenous (AV) access graft in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kei Kaneko, Study Director — W. L. Gore & Associates G.K
Locations (17):
- Japan (17):
  - Kaikoukai Central Clinic, Nagoya, Aichi-ken
  - Nagoya Vascular Access Clinic, Nagoya, Aichi-ken
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Kanazawa Cardiovascular Hospital, Kanazawa, Ishikawa-ken
  - Yokohama Dai-ichi Hospital, Yokohama, Kanagawa
  - Japanese Red Cross Kumamoto Hospital, Higashi, Kumamoto
  - Saitama Medical Center, Kawagoe, Saitama
  - Shizuoka General Hospital, Aoi, Shizuoka
  - Bouseidai1 Clinic, Numazu, Shizuoka
  - Haruguchi Vascular Access Clinic, Chiyoda City, Tokyo
  - Kichijoji Asahi Hospital, Musashino, Tokyo
  - Vascular Access Clinic Mejiro, Toshima City, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi
  - Fukuoka City Hospital, Fukuoka
  - Ikeda Vascular Access, Dialysis and Internal Medicine Clinic, Fukuoka
  - Osaka Vascular Access Temma Nakamura Clinic, Osaka

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GORE® VIABAHN® Stent Graft
Started | 124
Completed | 105
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 124
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.58 (5.39)
Smoking History [Count of Participants; unit: Participants]
  Currently Smoking | 9
  Past Smoking | 10
  No history of smoking | 35
  Unknown | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Loss of Primary Patency of Target Lesion
Description: Primary patency of target lesion is defined as the period during the patency was maintained from initial treatment until occlusion of target lesion or re-treatment of target lesion.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 124
Participants | 81

2. Primary Outcome: Number of Subjects With Loss of Secondary Patency of Target Lesion
Description: Secondary patency of target lesion is defined as the period during the patency was maintained from initial treatment (including the period of patency after re-treatment).
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 124
Participants | 17

3. Primary Outcome: Number of Subjects With Loss of Primary Patency of Vascular Access Circuit
Description: Primary patency of vascular access circuit is defined as the period during the patency was maintained from initial treatment until occlusion in vascular access or re-treatment in vascular access circuit.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 124
Participants | 98

4. Primary Outcome: Number of Subjects With Loss of Secondary Patency of Vascular Access Circuit
Description: Secondary patency of vascular access circuit is defined as the period during the patency was maintained from initial treatment until discontinuation of the use of vascular access circuit.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 124
Participants | 18

5. Primary Outcome: Mean Cumulative Number of Re-treatment Per Target Lesion
Description: Mean cumulative number of re-treatment in target lesion is defined as the number of re-treatment performed for target lesion after the initial treatment.
Time Frame: at 24 months
Population: number of target lesions evaluable at 24 months
Measure: Mean (95% Confidence Interval); unit: reinterventions per target lesion
Units Other Than Participants: lesions
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 90
Number analyzed (lesions) | 92
reinterventions per target lesion | 2.052 [1.601 to 2.502]

6. Primary Outcome: Number of Subjects Achieving Technical Success
Description: Technical Success is defined as < 30% residual stenosis after initial treatment.
Time Frame: Day 1
Population: Evaluable subjects. Technical success could not be determined among 14 subjects not assessed for residual stenosis.
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 110
Participants | 110

7. Primary Outcome: Number of Subjects Achieving Clinical Success
Description: Clinical Success is defined as the resumption of normal dialysis for at least one session after the initial treatment.
Time Frame: Day 1 to Month 1 follow up
Population: Number of subjects with 1 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 72
Participants | 72

8. Primary Outcome: Number of Subjects Experiencing Device and Procedure-related Adverse Events
Description: An adverse event (AE) is defined as any unfavorable or unintended sign (including abnormal laboratory changes), symptom, or illness associated with the use of a medical device. Unless worsening of severity or increasing of incidence during the surveillance, the primary disease of the patient is not considered an adverse event.
Time Frame: Day 1 to Month 1 follow up
Population: subjects on study at 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 122
Participants | 4

9. Primary Outcome: Number of Subjects Experiencing Device Defects
Description: A device defect is defined as a defect such as damage, malfunction, etc. that are widely unfavorable. Regardless of whether they are due to design, marketing, distribution, or use.
Time Frame: Day 1 to Month 1 follow up
Population: Subjects on study at 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | GORE® VIABAHN® Stent Graft
Number analyzed (Participants) | 122
Participants | 0

ADVERSE EVENTS:
Time Frame: Through 24 months (day 821)
Arm/Group | GORE® VIABAHN® Stent Graft
All-Cause Mortality (participants affected / at risk) | 19/124
Serious Adverse Events (participants affected / at risk) | 55/124
Other Adverse Events (participants affected / at risk) | 74/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® VIABAHN® Stent Graft (N=124)
Cardiac failure (Cardiac disorders) | 5 (5)
Myocardial infarction (Cardiac disorders) | 1 (1)
Artificial blood vessel occlusion (General disorders) | 5 (5)
Death (General disorders) | 5 (5)
Vascular stent occlusion (General disorders) | 20 (41)
Vascular stent stenosis (General disorders) | 6 (9)
Contrast media allergy (Immune system disorders) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 1 (1)
Infective spondylitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Shunt infection (Infections and infestations) | 3 (5)
Arteriovenous graft site pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 3 (5)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Diabetic macroangiopathy (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Subclavian vein stenosis (Vascular disorders) | 1 (3)
Venous occlusion (Vascular disorders) | 1 (1)
Venous stenosis (Vascular disorders) | 4 (13)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GORE® VIABAHN® Stent Graft (N=124)
Vascular stent occlusion (General disorders) | 39 (84)
Vascular stent stenosis (General disorders) | 40 (98)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 21 (56)
Venous stenosis (Vascular disorders) | 17 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI is required to obtain written permission from the Sponsor prior to publish trial results.

DOCUMENTS (2):
  • Study Protocol (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT04429243/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT04429243/SAP_001.pdf